CLINICAL TRIAL: NCT04336371
Title: Exploratory Prospective of Experienced by Patients in the Surgery of Skin Cancers of the Face in Interventional Dermatology Department
Acronym: VECUCHIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2019/46
Record Dates: First submitted 2020-03-31; First posted 2020-04-07 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Skin Cancer Face; Surgical Incision
Keywords: surgical; act- quality of life
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Anxiety level: patient's psychological experience the anxiety level
  Interventions: Diagnostic Test: Self-administered questionnaires

INTERVENTIONS:
Diagnostic Test: Self-administered questionnaires — Self-administered questionnaires by the patient will be given during visits in the following order:the self-administered questionnaires concerning the announcement consultation will be completed by the patient after consultation waiting room; self-questionnaires will be given in just before the operation waiting room (D0) just before the suture removal points (J10) and just before the follow-up visit (M3).

SUMMARY:
Surgery is the first-line treatment of localized skin cancers. Knowledge on the patient's psychological experience is limited. Therefore, the psychological impact on patients before, during and after surgery can be underestimated. Moreover, the diagnosis of cancer disturbs the patient's entire life and the onset of anxiety disorders is frequent following this announcement.

DETAILED DESCRIPTION:
The main objective of the study is to explore patients' experience assessing anxiety before, during and away from surgery. The investigators will distinguish the anxiety related to the surgical act itself and the anxiety related to the announcement of the disease.

The secondary objective is to assess the impact of surgery on quality of life, self-image and aesthetic satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 year-old
* Skin cancer on the face ((malignant lentigo, basal cell carcinoma and squamous cell carcinoma) for which a surgical treatment is proposed and will be performed in the Dermatology unit of the University Hospital (CHU) de Bordeaux
* Surgical procedure under local anesthesia
* Patient affiliated to Health Insurance
* Patients will sign consent after reading the information sheet explaining the objectives of the study.

Exclusion Criteria:

* Patients not able to complete the self-assessment questionnaires (difficulties for understanding or reading)
* Patient for whom there was no pre-op consultation in the center
* Patient for whom follow-up will not be possible in the center (because of remoteness for example)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with skin cancer on the face ((malignant lentigo, basal cell carcinoma and squamous cell carcinoma) for which a surgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2020-05-28 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Assess the patient's psychological experience in terms of anxiety, cosmetics and social aspects of surgery | Day 1
  Self-assessment questionnaires will be given to the patient
Assess the patient's psychological experience in terms of anxiety, cosmetics and social aspects of surgery | Day 10
  Self-assessment questionnaires will be given to the patient
Assess the patient's psychological experience in terms of anxiety, cosmetics and social aspects of surgery | Month 3
  Self-assessment questionnaires will be given to the patient

CONTACTS AND LOCATIONS:
Overall Officials: Marie BEYLOT-BARRY, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Hôpital Saint-André - CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carr EC, Nicky Thomas V, Wilson-Barnet J. Patient experiences of anxiety, depression and acute pain after surgery: a longitudinal perspective. Int J Nurs Stud. 2005 Jul;42(5):521-30. doi: 10.1016/j.ijnurstu.2004.09.014. Epub 2004 Nov 25. PMID 15921983
- [Background] Matthias AT, Samarasekera DN. Preoperative anxiety in surgical patients - experience of a single unit. Acta Anaesthesiol Taiwan. 2012 Mar;50(1):3-6. doi: 10.1016/j.aat.2012.02.004. Epub 2012 Mar 30. PMID 22500906
- [Background] Caumo W, Schmidt AP, Schneider CN, Bergmann J, Iwamoto CW, Bandeira D, Ferreira MB. Risk factors for preoperative anxiety in adults. Acta Anaesthesiol Scand. 2001 Mar;45(3):298-307. doi: 10.1034/j.1399-6576.2001.045003298.x. PMID 11207465
- [Background] Reddi D, Curran N. Chronic pain after surgery: pathophysiology, risk factors and prevention. Postgrad Med J. 2014 Apr;90(1062):222-7; quiz 226. doi: 10.1136/postgradmedj-2013-132215. Epub 2014 Feb 26. PMID 24572639
- [Background] Kain ZN, Sevarino FB, Rinder C, Pincus S, Alexander GM, Ivy M, Heninger G. Preoperative anxiolysis and postoperative recovery in women undergoing abdominal hysterectomy. Anesthesiology. 2001 Mar;94(3):415-22. doi: 10.1097/00000542-200103000-00009. PMID 11374599
- [Background] Gaudry E, Vagg P, Spielberger CD. Validation of the State-Trait Distinction in Anxiety Research. Multivariate Behav Res. 1975 Jul 1;10(3):331-41. doi: 10.1207/s15327906mbr1003_6. PMID 26829634
- [Background] Kindler CH, Harms C, Amsler F, Ihde-Scholl T, Scheidegger D. The visual analog scale allows effective measurement of preoperative anxiety and detection of patients' anesthetic concerns. Anesth Analg. 2000 Mar;90(3):706-12. doi: 10.1097/00000539-200003000-00036. PMID 10702461
- [Background] Lee EH, Klassen AF, Cano SJ, Nehal KS, Pusic AL. FACE-Q Skin Cancer Module for measuring patient-reported outcomes following facial skin cancer surgery. Br J Dermatol. 2018 Jul;179(1):88-94. doi: 10.1111/bjd.16671. Epub 2018 May 23. PMID 29654700
- [Background] Lee EH, Klassen AF, Nehal KS, Cano SJ, Waters J, Pusic AL. A systematic review of patient-reported outcome instruments of nonmelanoma skin cancer in the dermatologic population. J Am Acad Dermatol. 2013 Aug;69(2):e59-67. doi: 10.1016/j.jaad.2012.09.017. Epub 2012 Oct 24. PMID 23102770
- [Background] Chernyshov PV, Lallas A, Tomas-Aragones L, Arenbergerova M, Samimi M, Manolache L, Svensson A, Marron SE, Sampogna F, Spillekom-vanKoulil S, Bewley A, Forsea AM, Jemec GB, Szepietowski JC, Augustin M, Finlay AY. Quality of life measurement in skin cancer patients: literature review and position paper of the European Academy of Dermatology and Venereology Task Forces on Quality of Life and Patient Oriented Outcomes, Melanoma and Non-Melanoma Skin Cancer. J Eur Acad Dermatol Venereol. 2019 May;33(5):816-827. doi: 10.1111/jdv.15487. Epub 2019 Apr 8. PMID 30963614
- [Background] Rhee JS, Matthews BA, Neuburg M, Smith TL, Burzynski M, Nattinger AB. Skin cancer and quality of life: assessment with the Dermatology Life Quality Index. Dermatol Surg. 2004 Apr;30(4 Pt 1):525-9. doi: 10.1111/j.1524-4725.2004.30169.x. PMID 15056143
- [Background] van de Kar AL, Corion LU, Smeulders MJ, Draaijers LJ, van der Horst CM, van Zuijlen PP. Reliable and feasible evaluation of linear scars by the Patient and Observer Scar Assessment Scale. Plast Reconstr Surg. 2005 Aug;116(2):514-22. doi: 10.1097/01.prs.0000172982.43599.d6. PMID 16079683